CLINICAL TRIAL: NCT02632669
Title: A Prospective Stage IIS Clinical Trial Evaluating Hemi-Ablative Low Dose Rate (LDR) Brachytherapy for Localised Prostate Cancer
Brief Title: Hemi-Ablative Prostate Brachytherapy
Acronym: HAPpy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Stephen Langley, Professor of Urology & Clinical Director Royal Surrey & St Luke's Cancer Centre, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R&D12oncn0015
Record Dates: First submitted 2015-11-16; First posted 2015-12-17 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Prostatic Neoplasms; Cancer of the Prostate
Keywords: Focal brachytherapy; Seed implant; Quality of life; Toxicity
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemigland focal LDR brachytherapy (Experimental): Hemigland focal LDR brachytherapy using permanent iodine 125 seed implantation
  Interventions: Radiation: Hemigland focal LDR brachytherapy

INTERVENTIONS:
Radiation: Hemigland focal LDR brachytherapy — The treatment is limited to the hemigland that has been diagnosed with unilateral low to intermediate risk prostate cancer by means of pre-treatment staging with mpMRI and transperineal template biopsy. The affected hemigland will be treated with iodine-125 to a prescription dose of 145Gy. Patients will be assessed at baseline and subsequently at 6 weeks, 3, 6, 9, 12,18, 24 months after treatment with PSA and EN2 measurements and validated questionnaires relating to erectile, urinary, and bowel function and general health related quality of life. mpMRI and transperineal template biopsy will be performed 24 months after treatment.

SUMMARY:
This clinical study will evaluate side effects, quality of life and cancer control in patients with prostate cancer diagnosed on only one side of the prostate gland.

The diagnosis of unilateral prostate cancer will be made by means of a prostate transperineal template biopsy (TTB) and multiparametric magnetic resonance imaging (mpMRI).

Patients will be treated with low dose rate brachytherapy, using permanent iodine seed implants.Treatment will be limited to the side of the gland where the cancer has been diagnosed and is therefore called "focal" brachytherapy.

Prostate brachytherapy is usually applied to the whole prostate gland. After whole gland prostate brachytherapy urinary, bowel and sexual function may be affected. In this focal approach, the side effects will be evaluated by means of patient questionnaires.These will be repeated at various intervals after treatment.The results will be compared to the same questionnaires responded by patients who have undergone whole gland brachytherapy.Therefore an assessment can be made whether focal therapy produces fewer side effects than whole gland brachytherapy.The observation period will last for two years after treatment. A biopsy and mpMRI will be repeated after two years to evaluate prostate cancer control.

DETAILED DESCRIPTION:
This is a pilot Stage IIS study to evaluate the feasibility of performing a larger multicentre trial.The HAPpy study is a prospective development study offering hemi ablative LDR brachytherapy to 34 men with histologically proven low or intermediate risk localised prostate adenocarcinoma which affects a single lobe of the prostate.The data obtained from these 34 patients will be compared to matched patients from a retrospective cohort of whole gland brachytherapy patients treated in the same institution.Precise mapping and characterisation of the disease will be established using mp-MRI (T2-weighted and DCE(gadolinium)) imaging and transperineal template biopsy (TTB). Only the lobes with disease (left or right half of the gland) will be treated provided that the contralateral side is free of disease. Patients will be followed for two years post treatment at which time a further mp-MRI and TTB will confirm disease control outcomes.

Focal therapy for prostate cancer is a new idea and is considered an experimental treatment which needs to be evaluated within carefully conducted clinical trials . Rather than investigating focal therapy in a strict sense where only known areas of disease are treated, a more conservative approach needs to be taken until more information can be obtained regarding the outcomes of changing treatment techniques. Hemi-ablative focal therapy is considered to be a low-risk treatment and investigations into the performance of the technique should provide a pathway for future investigations of less conservative methodologies. Hemi-ablative focal therapy treats half of the prostate gland with a treatment margin, effectively treating at least 50% of the whole gland with a prescription dose. In theory, this should lessen the side effects associated with radical treatment while still maintaining disease control.This type of treatment is only suitable for patients with unilateral disease.

An international group of experts was established to form a consensus on how to design and conduct an LDR focal brachytherapy program for clinical trials. The group's findings were published by Langley et al and a dosimetric modelling study by Al Qaisieh et al.

Focal hemi gland brachytherapy will be delivered by means of an adaptation of same real-time planning technique (denominated 4D Brachytherapy) used to deliver whole gland LDR prostate brachytherapy. Stranded iodine 125 sources are implanted on the periphery of the prostate gland and loose iodine 125 sources are implanted within the central volume of the gland. Because all planning and dosimetry are done in real-time, radiotherapy physics will be able to adhere to the strict planning protocols required for this study.

Treatment planning: For standard whole-gland treatment, the whole prostate gland is delineated to form the Planning Target Volume (PTV) and the V100 is planned such that it covers the entire PTV plus a 0.5cm margin. For hemi-ablative focal treatments, the prostate will be divided into half and a new HTV (called the HemiTreatment Volume) is outlined on the side of the prostate determined to have clinically significant disease. A treatment margin of 0.5cm is considered around the HTV, which is similar when planning whole-gland treatment. In this way, >95% of the HTV is aimed to receive 100% of the prescription dose (V100). The V150 is situated in a semi-horseshoe shape in order to spare the urethra from high doses of radiation.

Dose parameters to critical organs are as follows:-

HEMI PROSTATE:

Prescription Dose 145Gy V100 = >95% V150 = 50-60% D90 = 140 - 160 Gy

URETHRA:

V150 <15%

RECTUM:

D0.1cc <200 Gy

The trial design follows recommendations published by the Balliol Collaboration under the Idea, Development, Exploration, Assessment, Long-term follow-up (IDEAL) model for a surgical study.

Data Collection and Statistics

1. Sample Size- Pilot Study There are no published results available and this technique has not been trialed to determine its effectiveness in disease control and quality of life outcomes. As such, a preliminary study is necessary to determine efficacy and feasibility before a large, multi-centre trial can be performed where a significant number of patients can be recruited for appropriate statistical analysis.

   The trial site currently treats ~300 patients per year for whole-gland brachytherapy. Of these 300 patients, ~25% present with unilateral disease that is low and intermediate risk. Recruitment will be over 18 months, in which time 100 patients should be eligible for the HAPpy trial. We anticipate a 25% drop-out rate after mp- MRI and template prostate mapping (TPM) biopsy results and a further 25% drop-out due to refusal to participate. This means that ~50 patients should be available for recruitment into the study over an 18 month period. In order to assess a decrease in side-effects (based on quality of life (QoL)) data of at least 10%, 34 patients will be required for the study. This is comparing two independent groups (prospective hemi group versus retrospective whole-gland group) when using α = 5%, β = 10%, and σ = 20%.
2. Data collection The main research co-ordinator is a qualified and experienced data manager. Data will be collected in both paper and electronic form and the data will be stored in one place and backed up twice on two different servers. Data will be held according to the Data Protection Act 1998 and pseudo anonymised as necessary. Each participant will be given a study number and this will be used on all of their study records. The patient number will be known to the chief investigator, the research co-ordinator, and the research radiographer or nurse assigned to the study. Data will be kept in a secure manner in the research offices with access to named individuals from the study group only. The paper records will be kept for a minimum of 10 years after the end of the study. A research radiographer or nurse will be appointed at the time of trial commencement to ensure that the Quality of Life (QOL) questionnaires are completed at each follow-up visit as required by the trial protocol. The research radiographer or nurse is also responsible for ensuring that each patient in the trial has appropriate appointments set up for each treatment, scanning (mp-MRI, biopsy), and follow-up visit and the necessary information is collected at each visit under the protocol. All clinic visit information including questionnaires, scans, biopsy results, and blood results will be kept in study records.
3. Analysis Thirty-four patients will be examined in the HAPpy trial and with this small sample number, non-parametric analysis of the data will be the most suitable. Patients will be paired or matched according to their tumour staging and pathology, age, and baseline scores. The Mann-Whitney U test, the Wilcoxon test, as well as tests for normality (if appropriate) of the data will be performed to determine if there are differences in the trial groups. Analysis of variance will be performed if the data is appropriate to use in this manner.

   Data to be collected:- IPSS + QoL questionnaire = Numerical scores, time-points IIEF-5 QoL questionnaire = Numerical scores, time-points EORTC-QLQ-PR25 bowel symptoms questionnaire = Numerical scores, time-points Dosimetry Values for PTV and HTV = Numerical V100, V150, D90 = Numerical Dose to the Urethra (V150) = Numerical Dose to the Rectum (D0.1cc) = Numerical Pathology review of biopsies (all) Standard reporting, qualitative, ranked mm of core invaded = Numerical Biopsy % core invaded = Numerical Prostate-specific antigen (PSA) = Numerical, time-points EN2 = Numerical, time-points Gleason Score= Numerical Staging = Standard reporting, qualitative, ranked

   Outcomes will be reported as estimates with 95% confidence intervals using appropriate methods based on the type of data. For patient reported outcomes with available baseline measurements, a comparison will be made with baseline values using paired analyses. Logistic regression will be used to investigate associations with potential risk factors for histological failure, considering PSA and EN2, Gleason score, cancer core length involvement (mm and %), number and % of positive biopsies for any cancer on TTB, stage and risk group. Sensitivity and specificity (with 95% confidence intervals) will be estimated in considering the use of standard PSA kinetics and thresholds for identifying clinically significant cancer. Scores from the quality of life questionnaires will be used in multivariable cross-sectional and longitudinal regression analysis comparing the treatment groups.

   Dosimetric evaluation to the PTV, HTV, and structures (urethra, rectum,bladder) will be performed (ultrasound real-time planning and post-operative CT). The dosimetry will be correlated with QoL information and disease control outcomes.

   Results from the TTB will be compared with the mp-MRI scans to evaluate the efficacy of using mp-MRI for diagnosis of disease. Disease modelling in three dimensions may be performed if a suitable physicist can be found to perform such an analysis.

   EN2 and PSA evaluation over time will be examined using regression analysis and compared between the two trial arms.

   Biopsy and mp-MRI results at 2-years (disease control outcomes) will be compared with pre-treatment biopsy and mp-MRI data and correlated with QoL information and dosimetry.

   Thirty-four patients will be examined in the HAPpy trial and with this small sample number, non-parametric analysis of the data will be the most suitable. Patients will be paired or matched according to their tumour staging and pathology, age, and baseline scores. The Mann-Whitney U test, the Wilcoxon test, as well as tests for normality (if appropriate) of the data will be performed on the data to determine if there are differences in the trial groups. Analysis of variance will be performed if the data is appropriate to use in this manner.
4. Reporting of Results The data will be analysed and submitted for peer reviewed journals for publication as full manuscripts. Abstracts to conferences will also be submitted for poster or oral presentation. An interim analysis at 12 months using histological and imaging data will be performed once sufficient data are available.

Data collection and reporting of results will follow the guidelines outlined in CONSORT and STROBE for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. TRUS biopsy (if taken):

   unilateral disease only
2. Template biopsy (TTB):

   unilateral disease only, AND Gleason < 7 (either 3+4 or 4+3)
3. mp-MRI results: Disease must present as unilateral (left or right) only
4. Stage T1-T2bN0M0 disease, as determined by local guidelines *
5. Serum PSA < 15
6. Prostate volume < 50cc
7. Eligible for brachytherapy as outlined in local guidelines*
8. Life expectancy > 10 years

Exclusion Criteria:

1. Men who have had previous radiation therapy
2. Men who have had androgen suppression/hormone treatment within the previous 12 months for their prostate cancer
3. Men with evidence of metastatic disease or nodal disease outside the prostate on bone scan or cross-sectional imaging.

   * https://www.rcr.ac.uk/quality-assurance-practice-guidelines-transperineal-ldr-permanent-seed-brachytherapy-prostate-cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 31 (Actual)
Dates: Start 2012-07-06 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Treatment related Urinary toxicity (symptoms) as recorded by the IPSS questionnaire score. | 2 years
  The International Prostate Symptom Score (IPSS) validated questionnaire will be used to score urinary toxicity (symptoms) after hemigland focal brachytherapy. Scores (mild = 0 to 7; moderate = 8 to 19; severe = 20 to 35) will be obtained pre-treatment and the outcomes reported as the change in score at 6 weeks, 3, 6, 9, 12, 18 and 24 months after treatment.
Treatment related Quality of Life (QoL) due to urinary symptoms as recorded by the Quality of Life (QoL) component of the IPSS questionnaire score. | 2 years
  The QoL component of the IPSS questionnaire will be used to score QoL due to urinary symptoms that may arise after hemigland focal brachytherapy. Scores (good = 0 to 2 ; acceptable = 3 to 4 ; poor = 5 to 6) will be obtained pre-treatment and the outcomes reported as the change in score at 6 weeks, 3, 6, 9, 12, 18 and 24 months after treatment.
Treatment related bowel toxicity (symptoms) as recorded by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life (QoL) questionnaire (30 PR 25) score. | 2 years
  The EORTC-QLQ-PR25 questionnaire will be used to score bowel toxicity (symptoms) after hemigland focal brachytherapy. Scores (normal bowel function = 4; mild bowel toxicity = 5 to 8 ; moderate toxicity = 9 to 12 ; severe toxicity = 13 to 16) will be obtained pre-treatment and the outcomes reported as the change in score at 6 weeks, 3, 6, 9, 12, 18 and 24 months after treatment.
Treatment related adverse events on Erectile function as recorded by the International Index of Erectile Function 5 (IIEF 5) questionnaire score. | 2 years
  The IIEF 5 validated questionnaire will be used to score erectile function after hemigland focal brachytherapy. Scores (no erectile dysfunction (ED) = 22 to 25; mild ED = 17 to 21; mild to moderate ED = 12 to 16; moderate ED = 8 to 11; severe ED = 5 to 7) will be obtained pre-treatment and the outcomes reported as the change in score at 6 weeks, 3, 6, 9,12,18 and 24 months after treatment.

SECONDARY OUTCOMES:
To evaluate tumor control of hemigland focal brachytherapy | 2 years
  The absence of clinically significant cancer in either treated or untreated prostate hemigland will be determined by Gleason score of transperineal template biopsy cores together with PI-RADS score of MRI imaging (T2, DWI and DCE) at two years after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Langley, MD, Principal Investigator — Royal Surrey NHS Foundation Trust
Locations (1):
- Royal Surrey NHS Foundation Trust, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahmed HU, Pendse D, Illing R, Allen C, van der Meulen JH, Emberton M. Will focal therapy become a standard of care for men with localized prostate cancer? Nat Clin Pract Oncol. 2007 Nov;4(11):632-42. doi: 10.1038/ncponc0959. PMID 17965641
- [Background] Eggener SE, Scardino PT, Carroll PR, Zelefsky MJ, Sartor O, Hricak H, Wheeler TM, Fine SW, Trachtenberg J, Rubin MA, Ohori M, Kuroiwa K, Rossignol M, Abenhaim L; International Task Force on Prostate Cancer and the Focal Lesion Paradigm. Focal therapy for localized prostate cancer: a critical appraisal of rationale and modalities. J Urol. 2007 Dec;178(6):2260-7. doi: 10.1016/j.juro.2007.08.072. Epub 2007 Oct 15. PMID 17936815
- [Background] Langley S, Ahmed HU, Al-Qaisieh B, Bostwick D, Dickinson L, Veiga FG, Grimm P, Machtens S, Guedea F, Emberton M. Report of a consensus meeting on focal low dose rate brachytherapy for prostate cancer. BJU Int. 2012 Feb;109 Suppl 1:7-16. doi: 10.1111/j.1464-410X.2011.10825.x. PMID 22239224
- [Background] Al-Qaisieh B, Mason J, Bownes P, Henry A, Dickinson L, Ahmed HU, Emberton M, Langley S. Dosimetry Modeling for Focal Low-Dose-Rate Prostate Brachytherapy. Int J Radiat Oncol Biol Phys. 2015 Jul 15;92(4):787-93. doi: 10.1016/j.ijrobp.2015.02.043. Epub 2015 Apr 28. PMID 25936808
- [Background] Langley SE, Laing RW. 4D Brachytherapy, a novel real-time prostate brachytherapy technique using stranded and loose seeds. BJU Int. 2012 Feb;109 Suppl 1:1-6. doi: 10.1111/j.1464-410X.2011.10824.x. PMID 22239223
- [Background] McCulloch P, Altman DG, Campbell WB, Flum DR, Glasziou P, Marshall JC, Nicholl J; Balliol Collaboration; Aronson JK, Barkun JS, Blazeby JM, Boutron IC, Campbell WB, Clavien PA, Cook JA, Ergina PL, Feldman LS, Flum DR, Maddern GJ, Nicholl J, Reeves BC, Seiler CM, Strasberg SM, Meakins JL, Ashby D, Black N, Bunker J, Burton M, Campbell M, Chalkidou K, Chalmers I, de Leval M, Deeks J, Ergina PL, Grant A, Gray M, Greenhalgh R, Jenicek M, Kehoe S, Lilford R, Littlejohns P, Loke Y, Madhock R, McPherson K, Meakins J, Rothwell P, Summerskill B, Taggart D, Tekkis P, Thompson M, Treasure T, Trohler U, Vandenbroucke J. No surgical innovation without evaluation: the IDEAL recommendations. Lancet. 2009 Sep 26;374(9695):1105-12. doi: 10.1016/S0140-6736(09)61116-8. PMID 19782876
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. PLoS Med. 2010 Mar 24;7(3):e1000251. doi: 10.1371/journal.pmed.1000251. PMID 20352064
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014 Dec;12(12):1495-9. doi: 10.1016/j.ijsu.2014.07.013. Epub 2014 Jul 18. PMID 25046131
- [Background] Barentsz JO, Weinreb JC, Verma S, Thoeny HC, Tempany CM, Shtern F, Padhani AR, Margolis D, Macura KJ, Haider MA, Cornud F, Choyke PL. Synopsis of the PI-RADS v2 Guidelines for Multiparametric Prostate Magnetic Resonance Imaging and Recommendations for Use. Eur Urol. 2016 Jan;69(1):41-9. doi: 10.1016/j.eururo.2015.08.038. Epub 2015 Sep 8. No abstract available. PMID 26361169
- [Result] Laing R, Franklin A, Uribe J, Horton A, Uribe-Lewis S, Langley S. Hemi-gland focal low dose rate prostate brachytherapy: An analysis of dosimetric outcomes. Radiother Oncol. 2016 Nov;121(2):310-315. doi: 10.1016/j.radonc.2016.09.014. Epub 2016 Nov 1. PMID 27814981
- [Result] Langley S, Uribe J, Uribe-Lewis S, Franklin A, Perna C, Horton A, Cunningham M, Higgins D, Deering C, Khaksar S, Laing R. Hemi-ablative low-dose-rate prostate brachytherapy for unilateral localised prostate cancer. BJU Int. 2020 Mar;125(3):383-390. doi: 10.1111/bju.14948. Epub 2019 Dec 23. PMID 31705700